CLINICAL TRIAL: NCT06852391
Title: JOULE - Metabolic Adaptation to Weight Loss in Response to a Behavioural Lifestyle Program With or Without Semaglutide in Adolescents With Obesity - a Randomized Controlled Trial
Brief Title: JOULE - Metabolic Adaptation to Weight Loss in Response to a Behavioural Lifestyle Program With or Without Semaglutide in Adolescents With Obesity
Acronym: JOULE-MARS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Diabetes Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18026
Record Dates: First submitted 2025-01-06; First posted 2025-02-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obesity (Disorder)
Keywords: Adaptive Thermogenesis; obesity; semaglutide; GLP-1 agonist; weight loss; Energy expenditure; Whole room calorimetry; MRI; MR elastography; Cold exposure; Liver stiffness; Brown adipose tissue; Pediatric; Quality of life
MeSH Terms: conditions — Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLP, then BLP+semaglutide (Active Comparator): Group A will engage in a BLP alone for the first six months of the study, then receive BLP and semaglutide (Wegovy®) for the last six months of the study, beginning with 0.25 mg subcutaneously weekly and being titrated every four weeks up to a maximum of 2.4 mg in approved doses 0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg.
  Interventions: Drug: Semaglutide Pen Injector; Behavioral: Behavioural Lifestyle Program (BLP)
- BLP and semaglutide (Experimental): In addition to BLP, Group B will receive semaglutide (Wegovy®) titrated to maximal dose tolerated, in approved doses of 0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg subcutaneously weekly for 6 months .
  Interventions: Drug: Semaglutide Pen Injector; Behavioral: Behavioural Lifestyle Program (BLP)

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Semaglutide will be delivered by a subcutaneous injection using an injectable pen once weekly. Semaglutide is formulated with 5 approved doses (0.25 mg, 0.5 mg, 1 mg, 1.7 mg, 2.4 mg). Treatment will commence with the lowest dose and will be increased every 4 weeks to the maximum tolerable dose where they will remain for the remainder of the treatment. Participants who are taking the drug will have monthly visits to assess any adverse events, dose titration and drug adherence.
  Other Names: Wegovy®
Behavioral: Behavioural Lifestyle Program (BLP) — The BLP will be delivered by the Growing Healthy Weight Management (GHWM) pediatric program at McMaster Children's Hospital. GHWM is a family-based program addressing health behaviours (nutritional pattern and eating behaviours, physical activity, sedentary time and sleep) and physical and mental health issues. In Year 1, the program typically includes 2 group sessions and monthly individualized sessions with the participant and their family. The interdisciplinary weight management team is comprised of a registered dietician, exercise physiologist, kinesiologist, social worker and/or psychologist, general pediatrician and pediatric endocrinologists.

SUMMARY:
The Joule MARS study is a single center, randomized, open label clinical trial aiming to explore the metabolic adaptations that occur in response to weight management in adolescents with obesity. Behavioural lifestyle intervention with and without a pharmacological intervention - semaglutide- will be studied. Study participants will be randomized to one of two groups. Group A will follow a behavioral lifestyle program (BLP) alone for 6 months, followed by BLP and treatment with semaglutide for six months. Group B will be enrolled in BLP and semaglutide from baseline to 6 months. The primary research question will assess, in youth aged 12-17 years diagnosed with obesity and enrolled in a weight management program, if the implementation of a BLP together with semaglutide, compared to the implementation of BLP alone for 6 months leads to less adaptive thermogenesis.

DETAILED DESCRIPTION:
The Joule MARS (Metabolic Adaptation to weight loss in Response to a behavioural lifestyle program with or without Semaglutide in adolescents with obesity) study is a single-center, randomized controlled trial designed to investigate the effects of a behaviour lifestyle program and the medication semaglutide on resting energy expenditure (REE), work efficiency during standard exercise on a cycle ergometer and related metabolic outcomes in adolescents with obesity. The study will involve two intervention groups:

Group A will participate in a behavioral lifestyle program (BLP) alone for 6 months followed by a combination of semaglutide treatment and a BLP for an additional 6 months.

Group B will receive semaglutide and a BLP for the first 6 months and then terminate the study.

The study objectives are to determine if, in youth aged 12-17 years with obesity and enrolled in a weight management program:

1. the implementation of a BLP and semaglutide, compared to the implementation of a BLP alone leads to less adaptive thermogenesis (AT) at 6 months;
2. the implementation of a BLP and semaglutide, compared to the implementation of a BLP alone for 6-month, leads to:

   Less increase in energy work efficiency during standardized exercise

   Differences in BAT activity

   Differences in health-related quality of life (HRQoL)
3. BLP and semaglutide, compared to BLP alone, lead to improvements in metabolic health measures (including lipids, glycemia, liver enzymes, hepatic fat and hepatic stiffness) after 6 months.
4. A longer time enrolled in BLP prior to addition of 6 months of semaglutide alters health outcome response to semaglutide.

A comprehensive assessment will be conducted throughout the study. Using whole-room indirect calorimetry, REE and muscle work efficiency, evaluated during standardized physical activity on a cycle ergometer, will be measured. Body composition (Dual energy x-ray absorptiometry and bioelectric impedance analysis), anthropometry (height, weight, waist circumference, BMI, BMI z score (WHO)), metabolic health, health related quality of life, hepatic fat and cold induced brown adipose tissue activity (MRI) will be assessed. Randomization will be managed via the REDCap EDC system.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 12-17 years
* Diagnosed with obesity (BMI ≥2 standard deviations above WHO Reference median)
* Enrolled in Growing Health Weight Management or Next Step pediatric clinics (ie. have at least one year of the program remaining).

Exclusion Criteria:

* Any contraindications for MRI (i.e. claustrophobia, implanted metal, metallic injuries recent tattoo or weight >300lb. Ineligible for imaging visit only.
* Use of atypical anti-psychotics.
* Use of the following medication classes: (i.e. Beta-blocker medications, Steatogenic medications, Anti-hyperglycemic medications, HIV drugs, Antidepressants, anxiolytic drugs, anti-psychotic drugs, Thyroid drugs, Antiemetic or amphetamine, dextromethorphan and metoclopramide.)
* Elevated alanine aminotransferase (ALT) > 5 x upper range of normal at screening.
* Use of glucose lowering or any anti-obesity medication in the previous 3 months.
* Known monogenic, syndromic or hypothalamic causes of obesity.
* Diagnosis of type 1 or 2 diabetes mellitus.
* Prior bariatric surgery or liver transplantation.
* Alcohol intake exceeding 3 drinks per week or reported cannabis use.
* Recent history of cigarette smoking (previous 3 months) - ineligible for imaging only.
* History or family history of multiple endocrine neoplasia 2 or medullary thyroid cancer.
* History of pancreatitis.
* Presence of untreated endocrine disorder.
* History of an eating disorder and / or history of suicidal ideation
* History of a cardiac condition that precludes exercise testing or unable to have exercise testing done in the GHWM pediatric clinic, inability to use a cycle ergometer.

Participant who does not have a peak power value obtained in the GHWM pediatric clinic

Female who is pregnant, breast-feeding or intends to become pregnant.

Female who refuses to use a means of contraception if sexually active.

Participation in any interventional clinical study within 90 days before screening.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Adaptive thermogenesis | 6, 12 months
  Adaptive thermogenesis will be calculated as the difference between measured and predicted REE after the intervention. Measured REE will be assessed with the participant awake, but at rest, in a whole room indirect calorimeter. Predicted REE will be calculated based on an equation derived using baseline data from this study population as is currently recommended. Variables that will be considered in deriving the equation include fat-free mass, fat mass, age and sex. We will compare adaptive thermogenesis (primary outcome) and work efficiency between the two treatments utilizing linear regression analysis. Separate analyses for males and females will ensure relevance of study findings to both sexes.

SECONDARY OUTCOMES:
Changes in energy work efficiency from baseline during standardized exercise | Baseline, 6, 12 months
  Energy work efficiency will be measured by measuring the physical activity energy expenditure (PAEE) from cycle ergometry using whole room calorimetry. This will be calculated as follows: Net mechanical efficiency (mechanical efficiency above resting): Ratio of power generated (kcal/min) / (PA EE - REE). One kcal/hour = 1.163 W Thus, [Power (W) x 0.01433 (kcal/min) / (PA EE (kcal/min) - resEE (kcal/min))] x100 = Work efficiency (%)
Brown Adipose Tissue (BAT) activity | From enrollment to 6 months and to 12 months
  Relative decline in supraclavicular fat proton density fat fraction after cold exposure as previously published (Ahmed et al., 2021)
Health-related quality of life (HRQoL) | Baseline to 6 months and to 12 months
  This will be measured using the Impact of Weight on Quality of Life kids (IWQOL-kids) questionnaire. Score ranges from 0 to 100, with 100 representing the best quality of life. In addition to a total score, there are scores on four domains:
  Physical Comfort (6 items)
  Body Esteem (9 items)
  Social life (6 items)
  Family Relations (6 items)
Total body mass, fat mass and lean mass | Baseline, 6, 12 months
  Body composition will be preferentially measured using Dual-energy X-ray absorptiometry (DXA) scans (Lunar PRODIGY Advance 8743; GE, Healthcare, Waukesha, WI). If the participant has a weight exceeding the limits for the machine, Bioelectrical Impedance Analysis (BIA) (InBody 570) will be utilized.
Hepatic fat content | Baseline, 6, 12 months
  Hepatic fat content will be measured via MRI conducted by a technician at St. Joseph's hospital at baseline, 6 months and 12 months using standardized techniques for precision, accuracy and determination of proton density fat fraction (PDFF) quantification of the whole liver
Hepatic stiffness | Baseline, 6 and 12 months
  Hepatic stiffness, an indicator of hepatic fibrosis, will be measured via Magnetic resonance elastography (MRE) using standardized techniques for precision and accuracy.
Fasting lipid profile | Baseline, 6, 12 months
  Differences in fasting lipids will be collected via fasting bloodwork. The types of lipids that will be collected will be triglycerides, cholesterol, High-density lipoprotein (HDL) and Low-density lipoprotein (LDL) (mmol/L).
Fasting insulin | Baseline, 6, 12 months
  Fasting insulin will be measured with bloodwork collected. HOMA-IR will be calculated to determine insulin resistance
Hemoglobin A1C | Baseline, 6 and 12 months
  Hemoglobin A1C to be measured in laboratory at Hamilton Health Sciences
Alanine aminotransferase | Baseline, 3, 6, 9 and 12 months
  ALT will be measured in the laboratory at Hamilton Health Sciences

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Morrison, MD FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided